CLINICAL TRIAL: NCT03436550
Title: Assessment of Portal Hypertension With Multiparametric MRI
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bachir Taouli, Professor of Radiology, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 16-1307; 1R01DK113272-01A1 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Portal Hypertension; Clinically Significant Portal Hypertension
Keywords: Hepatic Venous Pressure Gradient; Magnetic Resonance Imaging; Acoustic Radiation Force Impulse; Elastography; Ultrasound; Liver Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Chronic Liver Disease
  Interventions: Procedure: mpMRI; Procedure: ARFI US
- Control Group

INTERVENTIONS:
Procedure: mpMRI — Multiparametric MRI
  Groups: Patients with Chronic Liver Disease
Procedure: ARFI US — Acoustic radiation force impulse is a type of ultrasound elastography
  Groups: Patients with Chronic Liver Disease

SUMMARY:
The purpose of this study is to determine whether new multiparametric magnetic resonance imaging (MRI) methods (including diffusion-weighted MRI, dynamic contrast-enhanced MRI, MR elastography and phase-contrast imaging) can be useful in assessing liver damage and degree of portal hypertension (a complication of advanced liver fibrosis and cirrhosis) secondary to chronic liver disease, compared to ultrasound measurement of liver stiffness [acoustic radiation force impulse (ARFI) ultrasound] and routine blood tests. MRI uses magnetic fields to look at soft tissues in the body. This study will ultimately help to determine whether these methods will be useful in identifying liver disease and their complications that cannot be well-understood using current liver MRI techniques.

DETAILED DESCRIPTION:
Liver cirrhosis has been historically classified as a single histopathologic entity, as it is considered to be the latest fibrosis stage; however it is well known that cirrhosis encompasses different degrees of clinical severity. Advanced liver fibrosis and cirrhosis are commonly associated with portal hypertension, which is due to increased hemodynamic resistance of the liver leading to an increase in portal venous pressure. Portal hypertension leads to the development of esophageal varices associated with a high risk of bleeding, ascites and renal dysfunction. The definite diagnosis of portal hypertension is based on the measurement hepatic venous pressure gradient (HVPG), which is an indirect measure of portal pressure. This technique is invasive and not widely available. Portal hypertension may also be associated with a decrease in portal venous flow/velocity due to a higher parenchymal resistance to flow, and an increase in hepatic arterial flow secondary to an arterial buffer response that can be measured with phase-contrast magnetic resonance imaging (MRI). According to the researcher's recent data, the increased vascular pressure observed in portal hypertension affects liver and spleen stiffness as well as other viscoelastic properties measured with advanced 3D MR elastography, which may potentially be used as biomarkers of portal hypertension.

In this proposal, the researchers would like to validate noninvasive imaging biomarkers based on a short multiparametric MRI protocol for the quantification of changes in viscoelastic properties and flow metrics in the liver and spleen in relation to portal hypertension. This protocol could potentially be integrated in routine clinical MRI exams, and could significantly reduce the cost of care by decreasing the need for HVPG measurement, upper gastrointestinal endoscopies, and could provide a novel risk stratification scoring system of liver disease and portal hypertension based on MRI. This will be a highly significant progression in patients with liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease (including all etiologies of liver disease)
* 18 years of age and older
* Patient is able to give informed consent for this study
* Patients preferably (but not necessarily) underwent/will undergo:

  1. Liver biopsy (percutaneous or transjugular or surgical) performed within 6 months, as part of routine clinical care and/or HVPG measurement as part of their clinical care (within 6 months) and/or clinically indicated upper gastrointestinal endoscopy.

     and/or
  2. Liver transplant or liver resection performed as part of routine clinical care and/or
  3. Medical therapy for portal hypertension or TIPS placement as part of routine clinical care.

Control group

* Healthy volunteers without history of liver disease (will be used for the purpose of image optimization). These subjects will NOT undergo HVPG measurement.
* 18 years of age and older

Exclusion Criteria:

* Age less than 18 years
* Unable or unwilling to give informed consent
* Contra-indications to MRI

  1. Electrical implants such as cardiac pacemakers or perfusion pumps
  2. Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  3. Ferromagnetic objects such as jewelry or metal clips in clothing
  4. Pregnant subjects
  5. Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mount Sinai patients with concomitant portal pressure measurements and liver biopsy and/or upper GI endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Rate of diagnosis of portal hypertension (PH) | Within 12 months after initial index MRI
  Prospective diagnostic performance of mpMRI vs. ARFI US vs. routine serum markers for diagnosis of PH. Diagnosis of PH defined by HVPG ≥5 mmHg
Rate of diagnosis of clinically significant portal hypertension (CSPH) | Within 12 months after initial index MRI
  Prospective diagnostic performance of mpMRI vs. ARFI US vs. routine serum markers for diagnosis of CSPH. Diagnosis of CSPH (HVPG ≥10 mmHg)

SECONDARY OUTCOMES:
Rate of prediction of hepatic decompensation | Within 12 months of initial index MRI
  Prospective diagnostic performance of mpMRI and ARFI US for predicting hepatic decompensation. Rate of prediction of hepatic decompensation, defined as the occurrence of complications such as GI bleeding, encephalopathy, massive ascites (needing repeated paracentesis) or death.
Degree of ascites and TIPS patency | 3-6 months after TIPS procedure or beta-blockers have been prescribed
  Predicting response to TIPS (transjugular intrahepatic portosystemic shunt) and/or beta-blockers in patients with liver cirrhosis. Response will be defined on routine contrast-enhanced CT or MRI obtained within 3-6 months after TIPS or beta-blockers to establish the degree of ascites, and TIPS patency.

CONTACTS AND LOCATIONS:
Overall Officials: Bachir Taouli, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozkaya E, Bane O, Bhuiyan E, Geahchan A, Altinmakas E, Hectors SJ, Kennedy P, Abboud G, Pavuluri S, Ehman RL, Yin M, Lewis S, Bansal MB, Fischman A, Thung S, Schiano TD, Taouli B. Multiparametric MRI for Diagnosing Clinically Significant Portal Hypertension and Predicting Liver Decompensation. Liver Int. 2025 Nov;45(11):e70368. doi: 10.1111/liv.70368. PMID 41014103